CLINICAL TRIAL: NCT04256200
Title: Efficacy of Dienogest Versus Oral Contraceptive Pills on Pain Associated With Endometriosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Antoine Abou Moussa, Professor of Obstetrics and Gynecology/principal investigator, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OGY.AA.07
Record Dates: First submitted 2020-01-15; First posted 2020-02-05 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Endometriosis
Keywords: endometriosis; oral contraceptive pills; progestin
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Tablets; drospirenone and ethinyl estradiol combination; Contraceptives, Oral, Combined

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dienogest (Active Comparator): Deinogest (Visanne) 2mg/day orally for 24 weeks
  Interventions: Drug: Dienogest 2 MG Oral Tablet
- Oral Contraceptive Pills (Active Comparator): Oral contraceptive pill (Yasmin, 0.03mg Ethinyl Estradiol and 3mg Drospirenone) orally daily for 24 weeks
  Interventions: Drug: Yasmin

INTERVENTIONS:
Drug: Dienogest 2 MG Oral Tablet — Deinogest (Visanne) 2mg/day, orally for 24 weeks versus combined OCP (Yasmin, 0.03mg
  Other Names: Visanne
  Arms: Dienogest
Drug: Yasmin — 0.03mg Ethinyl Estradiol and 3mg Drospirenone daily for 24 weeks
  Other Names: combined oral contraceptive
  Arms: Oral Contraceptive Pills

SUMMARY:
Endometriosis is a chronic inflammatory disease, frequently associated with dysmenorrhea, dyspareunia and abdomino-pelvic pain limiting quality of life. Most medical therapies aim to alleviate the severity of symptoms. Recent guidelines recommend the use of either OCPs or progestins as a first-line treatment of pain associated with endometriosis. The effectiveness of both OCPs and dienogest, a fourth-generation progestin, for endometriosis treatment has been demonstrated. The literature is rich with data comparing the use of Visanne or OCPs to placebo or GnRH analogs. However, there are no head to head studies comparing their efficacy in the management of endometriosis associated pain. The study aims to evaluate if Dienogest (Visanne) is not inferior in efficacy to oral contraceptive pills (Yasmin) in controlling pain associated with endometriosis?

DETAILED DESCRIPTION:
Endometriosis is defined as the presence of endometrial tissue outside the uterus, which induces a chronic inflammatory reaction. It is an estrogen-dependent associated with pelvic pain and infertility. It is a relatively common chronic gynecological disease that affects approximately 10% of reproductive aged women. Patients with endometriosis often suffer from dysmenorrhea, dyspareunia, dysuria, and chronic abdominal or pelvic pain, resulting in a severely limited quality of life. The aim of most medical therapies is to alleviate the severity of symptoms. Commonly used hormonal therapies include combined oral contraceptives (OCP), progestogens, gonadotropin-releasing hormone (GnRH) agonists, androgens and antiprogestogens, all of which are considered to have similar efficacy but different tolerability profiles, which are often suboptimal. To date, the most widely used agent for the medical treatment of endometriosis is oral contraceptive (albeit off-label). In particular, evidence supporting the efficacy of estrogen-progestin therapy (EP) in pain control and reducing the risk of recurrence in women undergoing surgery for endometriosis. In recent years, the effectiveness of dienogest, a fourth-generation progestin, for endometriosis treatment has been demonstrated. Dienogest seems to be as effective as gonadotrophin-releasing hormone-a (GnRH-a) in terms of endometriosis-related pelvic pain improvement. The aim of this study is to evaluate the efficacy of Visanne versus OCP treatment of endometriosis associated pelvic pain in a double-blinded randomized controlled pilot study. It is a two armed pilot study; each group will include 50 patients. Women with endometriosis will be randomized to receive either DNG (n=50) or OCPs (n=50). The diagnosis of endometriosis will be by clinical evaluation, laparotomy, laparoscopy, or imaging analysis (combination of magnetic resonance imaging and ultrasonography) of endometriotic ovarian chocolate cysts.The first group will receive Deinogest (Visanne) 2mg/day, orally for 24 weeks. The second group will receive monophasic combined OCP (Yasmin, Ethinyl Estradiol and Drospirenone) daily for 24 weeks. The treating physician and the patients will be blinded to the treatment option. The relief of symptoms and efficacy will be evaluated by questionnaire on follow up visits at 3 and 6 month of the treatment. Data collected will be analyzed and compared between the 2 groups. We hypothesize that there will be no difference in pain scores, efficacy and safety between the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed or suspected of endometriosis on clinical evaluation (VAS score more than 5 and presence of subjective symptoms), surgical or imaging studies, and not taking any pain killer or other hormonal treatment for the moment
* Age 20-45
* Regular menstrual cycles
* The presence of subjective symptoms during menstruation (at least one from among lower abdominal pain, lumbago, defecation pain, nausea, and headache)
* The presence of subjective symptoms during non-menstruation (at least one from among lower abdominal pain, lumbago, defecation pain, dyspareunia, and pain on internal examination).

Exclusion Criteria:

* Undiagnosed genital bleeding
* Use of any hormonal therapy for endometriosis within 16 weeks before enrollment
* A history of severe adverse drug reactions or hypersensitivity to steroid hormone
* Having undergone surgery therapy or surgical examination for endometriosis within a menstrual cycle before the start of medication
* Previous failure of treatment with the OCP used in the current study
* Contraindications to OCP or Dienogest use
* Smokers >35
* A history or complication of thrombosis/embolism
* Migraines with aura
* Depression
* Patients on anti-epileptics
* Diabetes Mellitus with vascular involvement
* Liver diseases
* Known or suspected sex hormone dependent malignancies
* Repeat surgery for endometriosis
* Patient consulting for infertility
* Pregnant or nursing
* Planning for pregnancy in near future.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2017-02-07 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Endometriosis-associated pelvic pain | 6 months
  be the absolute change in endometriosis -associated pelvic pain from baseline to end of treatment, assessed by the Visual Analogue Scale (VAS): with "absence of pain" corresponding to the value "0" and "unbearable pain" corresponding to the value "10"

SECONDARY OUTCOMES:
Impact on Quality of life | 6 months
  Outcome quality of life will be assessed using Endometriosis Health Profile 30 (EHP30) with each item of this questionnaire can be answered by choosing one of the following (Never, rarely,sometimes, often and always). The endometriosis health profile is a patient-generated questionnaire in which the items were developed from interviews with women with the condition ( Obtained from Oxford University Press) .
incidence of side effects | 6 months
  Incidence of possible side effects including headache, migraine,nausea, vomiting, abdominal pain/discomfort, breast pain or tenderness, mood swings, premenstrual syndrome, decreased libido, fatigue, weight changes and menstrual irregularities
Patient Tolerability | 6 months
  Assessing tolerability to side effects via numerical scale from zero to ten ( zero not bothersome at all , ten maximum possible)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Abu Musa, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Derived] El Taha L, Abu Musa A, Khalifeh D, Khalil A, Abbasi S, Nassif J. Efficacy of dienogest vs combined oral contraceptive on pain associated with endometriosis: Randomized clinical trial. Eur J Obstet Gynecol Reprod Biol. 2021 Dec;267:205-212. doi: 10.1016/j.ejogrb.2021.10.029. Epub 2021 Oct 30. PMID 34826668